CLINICAL TRIAL: NCT00842582
Title: Neoadjuvant Azacitidine With Carboplatin and Paclitaxel for Suboptimal Newly Diagnosed Ovarian Cancer
Brief Title: Azacitidine With Carboplatin and Paclitaxel for Newly Diagnosed Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No enrollment. Unable to recruit due to lack of eligible patients.
Sponsor: Loyola University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200777
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Ovarian Cancer
Keywords: Ovarian cancer; chemotherapy; azacitidine
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single group assignment (Experimental): Patients will receive Azacitidine at 20, 40, or 75 milligrams per meter squared subcutaneous once daily for 7 days.
  Interventions: Drug: Azacitidine

INTERVENTIONS:
Drug: Azacitidine — Azacitidine 20 milligrams per meter squared subcutaneous once daily for 7 days.
Drug: Azacitidine — Azacitidine 40 milligrams per meter squared subcutaneous once daily for 7 days.
Drug: Azacitidine — Azacitidine 75 milligrams per meter squared subcutaneous once daily for 7 days.

SUMMARY:
This is a clinical trial for women with newly diagnosed ovarian cancer. The purpose of this study is to determine if the addition of a drug called azacitidine (Vidaza®)when added to carboplatin and paclitaxel will change the genetic material of the tumor so that the chemotherapy drugs work better.

The study will also determine what the maximum tolerated dose of azacitidine that may be safely used in combination with carboplatin and paclitaxel.

DETAILED DESCRIPTION:
Ovarian cancer is a highly chemosensitive tumor with good responses to first line chemotherapy. The problem is the high rate of relapse, especially in advanced disease

Relapses are likely due to the presence of chemoresistant cells that escape from first line platinum and taxane based regimens. Therefore, outcomes may be improved by adding treatment to initial standard therapy that makes resistant cells sensitive to chemotherapy. There are multiple targeted pathways that may achieve this goal. One promising path is epigenetics.

The reasons for this trial are multifold. First, methylation pathways have been proven in tissue models to be integral to ovarian cancer pathogenesis. Second, cisplatin and azacitidine are synergistic, and therefore would be promising in combination to improve ovarian cancer outcomes by combating cisplatin resistance, which is a major cause of ovarian cancer mortality. It has been proven that azacitidine/decitabine reverses platinum resistance. Third, azacitidine has shown tolerable toxicity and promise in clinical trials to date. Ideally, ovarian cancer outcomes are likely to be improved by the addition of treatment that wipes out chemoresistant cells, thus preventing relapse.

This study is a phase I, non-randomized, dose escalation treatment study using azacitidine in combination with intravenous chemotherapy with Paclitaxel and carboplatin.

All patients will receive the chemotherapy drugs Carboplatin and Paclitaxel. Patients will then be randomized to receive one of three different doses of Azacitidine.

ELIGIBILITY:
Inclusion Criteria:

* Stage III or IV epithelial ovarian cancer, fallopian tube cancer, or primary peritoneal cancer
* Appropriately signed and documented informed consent form, with documentation of the informed consent process
* Age more than 18 years old
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Life expectancy greater than 12 months
* Adequate baseline bone marrow function: absolute neutrophils count greater than 1500 cells/microliter, platelet count greater than 100,000 cells per microliter
* Adequate liver function: bilirubin than 1.5 times the upper limit of normal. Higher levels of Bilirubin are acceptable if these can be attributed to active hemolysis or ineffective erythropoiesis. Serum glutamic-oxaloacetic transaminase (SGOT) (aspartate aminotransferase (AST)) or serum glutamic-pyruvic transaminase (SGPT) (alanine aminotransferase (ALT)) levels less than or equal 2 x Upper Limit of Normal (ULN).
* Adequate renal function: Serum creatinine levels less than or equal to 1.5 times ULN
* Patients must have ascites and be considered not candidates for upfront surgery because of disease bulk (not because of overall health).
* Women of childbearing potential must have a negative serum pregnancy test prior to azacitidine treatment.
* Women of childbearing potential should be advised to avoid becoming pregnant and men should be advised to not father a child while receiving treatment with azacitidine.

Exclusion Criteria:

* Ongoing serious infection
* Neuropathy greater than grade 2 at baseline
* Major surgery within 2 weeks prior to enrollment
* Concurrent investigational treatment, antineoplastic treatment, hormonal treatment, or radiation therapy
* Prior bone marrow transplant
* prior radiation to the pelvis
* radiation therapy for malignancy within the past 5 years
* Other malignancy within the past 5 years except non-melanoma skin cancer.
* Known or suspected hypersensitivity to azacitidine or mannitol
* Pregnant or breast feeding
* Patients with advanced malignant hepatic tumors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
The primary goal is to find the lowest dose of azacitidine combined with carboplatin and Paclitaxel, at which toxicity is reasonable, and methylation changes are clinically significant (at which there is a change in gene expression. | 15 days

SECONDARY OUTCOMES:
Secondary endpoints are disease free survival, overall survival, toxicity, quality of life as measured by the Functional Assessment of Cancer Therapy-Ovarian Cancer symptom (FOSI) index, and basic science correlate. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Laura Horvath, MD, Principal Investigator — Loyola University Cardinal Bernadin Cancer Center
Locations (2):
- United States (2):
  - Loyola Univeristy Medical Center, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - Central Dupage Hospital, Winfield, Illinois

IPD SHARING:
Plan to Share IPD: No